CLINICAL TRIAL: NCT00096044
Title: CC-5013 Alone or in Combination With Rituximab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Lenalidomide With or Without Rituximab in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000391767; RPCI-I-18103 (Other: Roswell Park Cancer Institute); CELGENE-RV-CLL-PI-005 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Lenalidomide (Experimental): Patients receive oral lenalidomide (CC-5013) once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: rituximab; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab — IV
Drug: lenalidomide — Oral

SUMMARY:
RATIONALE: Biological therapies such as lenalidomide use different ways to stimulate the immune system and stop cancer cells from growing. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining lenalidomide with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying the how well giving lenalidomide with or without rituximab works in treating patients with relapsed or refractory chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the best cytostatic response rate (including complete response, partial response, or stable disease) in patients with relapsed or refractory chronic lymphocytic leukemia treated with lenalidomide (CC-5013).

Secondary

* Determine the cytostatic response rate in patients who progress on CC-5013 and are then treated with CC-5013 and rituximab.
* Determine the safety of these regimens in these patients.
* Determine time to progression in patients treated with these regimens.

OUTLINE: This is an open-label, non-randomized, pilot study.

Patients receive oral lenalidomide (CC-5013) once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) receive 2 additional courses beyond CR.

Patients with disease progression receive oral CC-5013 once daily on days 1-21 and rituximab IV on days 1, 8, and 15 during the first treatment course and on days 1 and 15 of all subsequent courses. Treatment repeats every 28 days for up to 6 courses in the absence of further disease progression. Patients who achieve CR receive 2 additional courses beyond CR.

Patients are followed at 1 month and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL) by flow cytometry

  * Relapsed or refractory disease
* Measurable disease, defined by 1 of the following criteria:

  * Absolute lymphocyte count ≥ 5,000/mm^3
  * Measurable lymphadenopathy or organomegaly
* Received ≥ 1 prior therapy for CLL

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 30,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2 times upper limit of normal (ULN) (5 times ULN if hepatic metastases are present)

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method (including barrier) contraception during and for 3 months after study participation
* No known hypersensitivity to thalidomide
* No erythema nodosum characterized by a desquamating rash after prior thalidomide or similar drug administration
* No known anaphylaxis or immunoglobulin E-mediated hypersensitivity to murine proteins
* No serious medical condition or laboratory abnormality that would preclude study participation
* No psychiatric illness that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior lenalidomide (CC-5013)
* No concurrent thalidomide

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since prior therapy for CLL
* At least 28 days since prior experimental drug or therapy
* No other concurrent anticancer therapies
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lee, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Lenalidomide
Started | 45
Completed | 11
Not Completed | 34
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 21
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Oral Lenalidomide
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) on Single Agent CC-5013 at 6 Months
Description: Percentage of patients achieving CR, PR or maintaining SD using the 1996 NCI-WF Criteria. CR: absence of lymph nodes and constitutional symptoms; no hepatomegaly or splenomegaly by physical examination; neutrophil count >1500/μL; platelet count >100,000/μL; untransfused hemoglobin concentration >11.0g/dL; lymphocyte count <4000/μL; bone marrow sample must be at least normocellular for age; with less than 30% of nucleated cells being lymphocytes and no lymphoid nodules. PR: ≥50% decrease in lymphocyte count from baseline; ≥50% reduction in lymph nodes from baseline; ≥50% reduction in the size of the liver/spleen from baseline; neutrophil count ≥1500/μL or ≥50% improvement from baseline; platelet count ≥100,000/μL or ≥50% improvement from baseline; untransfused hemoglobin concentration ≥11.0g/dL or ≥50% improvement from baseline. Patients have not exhibited as reappearance of malignant CLL clone on flow cytometry or by PCR analysis in blood or bone marrow, are considered to have SD.
Time Frame: at 6 Months
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral Lenalidomide
Number analyzed (Participants) | 45
percentage of participants | 68.9 [53.4 to 81.8]

2. Secondary Outcome: Percentage of Patients Achieving a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) on Combination Therapy of CC-5013+Rituximab
Description: Percentage of patients achieving CR, PR or maintaining SD using the 1996 NCI-WF Criteria. CR: absence of lymph nodes and constitutional symptoms; no hepatomegaly or splenomegaly by physical examination; neutrophil count >1500/μL; platelet count >100,000/μL; untransfused hemoglobin concentration >11.0g/dL; lymphocyte count <4000/μL; bone marrow sample must be at least normocellular for age; with less than 30% of nucleated cells being lymphocytes and no lymphoid nodules. PR: ≥50% decrease in lymphocyte count from baseline; ≥50% reduction in lymph nodes from baseline; ≥50% reduction in the size of the liver/spleen from baseline; neutrophil count ≥1500/μL or ≥50% improvement from baseline; platelet count ≥100,000/μL or ≥50% improvement from baseline; untransfused hemoglobin concentration ≥11.0g/dL or ≥50% improvement from baseline. Patients who have not exhibited as reappearance of malignant CLL clone on flow cytometry or by PCR analysis in blood or bone marrow, are considered to have SD.
Time Frame: 5 years
Population: All treated with combination therapy of CC-5013+Rituximab and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral Lenalidomide
Number analyzed (Participants) | 8
percentage of participants | 100 [63.1 to 100]

3. Secondary Outcome: Number of Participants With Adverse Events on Single Agent CC-5013
Description: Number of Participants with Adverse Events on Single Agent CC-5013, Graded According to NCI CTCAE Version 3.0
  Please refer to the adverse event reporting for more detail.
Time Frame: 1 year
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Lenalidomide
Number analyzed (Participants) | 45
Participants
  Grade 1 | 0
  Grade 2 | 3
  Grade 3 | 7
  Grade 4 | 33
  Grade 5 | 2

4. Secondary Outcome: Number of Participants With Adverse Events on Combination Therapy of CC-5013+Rituximab
Description: Number of Participants with Adverse Events on Combination Therapy of CC-5013+Rituximab, Graded According to NCI CTCAE Version 3.0
Time Frame: Up to 30 days from last date of institution of combination therapy of CC-5013+Rituximab.
Population: All treated with combination therapy of CC-5013+Rituximab and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Lenalidomide
Number analyzed (Participants) | 8
Participants
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 3
  Grade 4 | 3

5. Secondary Outcome: Time to Progression for Single Agent CC-5013
Description: Progressive disease is defined as reappearance of malignant CLL clone on flow cytometry or by PCR analysis in blood or bone marrow using the 1996 NCI-WF Criteria.
Time Frame: 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oral Lenalidomide
Number analyzed (Participants) | 45
months | 23.0 [12.1 to 78.7]

6. Secondary Outcome: Time to Progression for the Combination Therapy of CC-5013+Rituximab
Description: as for outcome 5
Time Frame: Every month up to 6 months and every 3 months thereafter up to 5 years
Population: All treated with combination therapy of CC-5013+Rituximab and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oral Lenalidomide
Number analyzed (Participants) | 8
months | 18.7 [0.9 to 23.0]

ADVERSE EVENTS:
Arm/Group | Oral Lenalidomide
Serious Adverse Events (participants affected / at risk) | 29/45
Other Adverse Events (participants affected / at risk) | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Lenalidomide (N=45)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (16)
Neutropenia (Blood and lymphatic system disorders) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (3)
Lobar pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 12 (15)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Intestinal anastomosis (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Lenalidomide (N=45)
Anaemia (Blood and lymphatic system disorders) | 35 (51)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 20 (44)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 41 (128)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 41 (79)
Bradycardia (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardiac flutter (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Cataract (Eye disorders) | 2 (2)
Eye irritation (Eye disorders) | 1 (1)
Eye oedema (Eye disorders) | 2 (2)
Lacrimation increased (Eye disorders) | 3 (3)
Ocular hyperaemia (Eye disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (2)
Photopsia (Eye disorders) | 1 (1)
Scleral discolouration (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 6 (7)
Visual impairment (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 11 (13)
Abdominal pain (Gastrointestinal disorders) | 10 (12)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 24 (44)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Eructation (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (17)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2)
Painful defaecation (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (12)
Asthenia (General disorders) | 23 (28)
Axillary pain (General disorders) | 1 (1)
Chest pain (General disorders) | 5 (7)
Chills (General disorders) | 1 (1)
Crepitations (General disorders) | 2 (2)
Early satiety (General disorders) | 1 (1)
Effusion (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 43 (70)
Feeling abnormal (General disorders) | 1 (1)
Feeling hot (General disorders) | 2 (2)
Influenza like illness (General disorders) | 4 (4)
Irritability (General disorders) | 1 (1)
Local swelling (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Oedema (General disorders) | 11 (13)
Oedema peripheral (General disorders) | 16 (26)
Pain (General disorders) | 3 (5)
Pyrexia (General disorders) | 16 (18)
Tenderness (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 11 (19)
Jaundice (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Clostridial infection (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Eye infection staphylococcal (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 4 (4)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Herpes zoster disseminated (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (6)
Opportunistic infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 5 (6)
Respiratory tract infection (Infections and infestations) | 3 (4)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 10 (18)
Tooth abscess (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 12 (35)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 9 (10)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Splenosis (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 14 (27)
Aspartate aminotransferase (Investigations) | 1 (1)
Aspartate aminotransferase decreased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 15 (26)
Blood alkaline phosphatase increased (Investigations) | 18 (18)
Blood bilirubin increased (Investigations) | 3 (5)
Blood creatine decreased (Investigations) | 2 (2)
Blood creatinine (Investigations) | 4 (4)
Blood creatinine decreased (Investigations) | 3 (3)
Blood creatinine increased (Investigations) | 3 (5)
Blood glucose increased (Investigations) | 1 (1)
Blood phosphorus (Investigations) | 4 (4)
Blood phosphorus decreased (Investigations) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood urea decreased (Investigations) | 4 (4)
Blood urea increased (Investigations) | 15 (15)
Blood uric acid decreased (Investigations) | 5 (5)
Blood uric acid increased (Investigations) | 3 (3)
Breath sounds abnormal (Investigations) | 2 (2)
Immunoglobulins decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (3)
Protein total decreased (Investigations) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (3)
Troponin (Investigations) | 1 (1)
Weight decreased (Investigations) | 13 (15)
Weight increased (Investigations) | 1 (1)
pH urine abnormal (Investigations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 17 (19)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (16)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (14)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 7 (7)
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 (7)
Hyperproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 (31)
Hypocalcaemia (Metabolism and nutrition disorders) | 27 (43)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 20 (22)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5)
Hypoproteinaemia (Metabolism and nutrition disorders) | 21 (21)
Hypouricaemia (Metabolism and nutrition disorders) | 3 (4)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (19)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 29 (35)
Burning sensation (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 2 (3)
Dizziness (Nervous system disorders) | 16 (23)
Headache (Nervous system disorders) | 14 (17)
Hypoaesthesia (Nervous system disorders) | 5 (6)
Lethargy (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 3 (3)
Migraine with aura (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 12 (13)
Paraesthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (3)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 4 (5)
Disorientation (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9)
Mood altered (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urethral spasm (Renal and urinary disorders) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (30)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (34)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 12 (16)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (15)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 27 (40)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 7 (8)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 7 (8)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Glaucoma drug therapy (Surgical and medical procedures) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1)
Tooth repair (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Lymphoedema (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes